CLINICAL TRIAL: NCT04285554
Title: A Prospective, Single-Arm, Multi-Center Study of the Metavention Integrated Radio Frequency Denervation System to Improve Glycemic Control in Type 2 Diabetic Subjects
Brief Title: Evaluation of the Integrated Radio Frequency Denervation System to Improve Glycemic Control in Type 2 Diabetic Subjects
Acronym: DeLIVER
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Metavention (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Device Feasibility
Other Study IDs: 932
Record Dates: First submitted 2020-02-19; First posted 2020-02-26 (Actual); Last update posted 2023-03-15 (Actual); Status verified 2023-03

CONDITIONS: Diabetes Mellitus, Type 2
Keywords: Metabolic Syndrome; NAFLD; Hypertension; High Blood Pressure; Glycemic Control; Diabetes; Denervation; Sympathetic Nervous System
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Metabolic Syndrome; Non-alcoholic Fatty Liver Disease; Hypertension; Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: The study is a prospective, single-arm, multi-center, non-randomized trial
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes

ARMS (1):
- Hepatic Denervation (Experimental)
  Interventions: Device: iRF System Hepatic Denervation

INTERVENTIONS:
Device: iRF System Hepatic Denervation — The iRF System is a percutaneous, catheter-based device which uses RF energy to circumferentially denervate the sympathetic nerves surrounding the common hepatic artery (CHA).

SUMMARY:
The objective of this early feasibility study is to evaluate the safety and performance of intravascular hepatic denervation using the Metavention Integrated Radio Frequency Denervation System (iRF System) to improve glycemic control in type 2 diabetes subjects.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥22 and ≤70 years old
2. Type 2 diabetes diagnosis meeting the following criteria:

   1. HbA1c > 7.0% and ≤ 9.0% (53 mmol/mol - 75 mmol/mol), AND
   2. On at least two anti-diabetic medications; one at the highest tolerated dose with no changes in medication dose in the 12 weeks prior to the first screening visit
3. Waist circumference ≥102 cm (male) and ≥88cm (female)
4. Diagnosis of hypertension: SBP ≥140mmHg OR SBP ≥130mmHg on hypertension medication(s)
5. Documented status of stable lifestyle modifications
6. Women of childbearing potential (WOCBP) must be using at least one acceptable method of contraception throughout the study

Exclusion Criteria:

1. BMI >40 kg/m2
2. Diagnosis of type 1 diabetes
3. Use of insulin within 90 days of consent
4. Two or more self-reported or documented severe hypoglycemia events (severe hypoglycemia event defined as: hypoglycemia associated with severe cognitive impairment requiring external assistance for recovery) in the 180 days prior to Index Procedure
5. One or more documented hyperglycemia episodes requiring hospitalization in the 180-days prior to Index Procedure
6. During medication run in period, uncontrolled hyperglycemia noted by a fasting glucose value of >270mg/dL or >360mg/dL at any point that is then confirmed by a second measurement (not on the same day)
7. A history of bariatric surgery, renal denervation, baroreflex activation therapy, or liver transplant, or these procedures are planned in the 365 days following Index Procedure
8. Any surgical procedure within 30 days prior to Index Procedure
9. History of or current symptomatic gallstones (e.g., cholecystitis, bile duct dilatation) without a cholecystectomy being performed (Note: subjects who have had a cholecystectomy are not excluded)
10. Previous hepatobiliary surgery/intervention that in the opinion of the investigator could preclude the ability to perform denervation of the common hepatic artery
11. Currently taking the following medications within 90 days prior to screening and/or there is a need or anticipated need for these medications during the study:

    1. Systemic corticosteroids
    2. Anticonvulsants
    3. Centrally acting sympatholytics
12. Use of anticoagulation therapy which cannot be discontinued from 7 days before to 14 days after the Index Procedure
13. Any other condition(s) that would compromise the safety of the Subject or compromise study quality as judged by the Investigator
14. eGFR <45 mL/min/1.73 m2
15. History or diagnosis of proliferative retinopathy or advanced autonomic neuropathy (e.g., orthostatic hypotension attributable to autonomic neuropathy, a diagnosis of gastroparesis, or a clinical history strongly suggestive of delayed gastric emptying)
16. Myocardial infarction, unstable angina within 1 year prior to consent
17. Widespread atherosclerosis with documented intravascular thrombosis or unstable plaques
18. Documented history or concurrent signs of significant thyroid disease NOTE: If a subject is on chronic thyroid drug treatment, and has a serum TSH test result in normal range at Screening they may enter study
19. Uncorrectable bleeding diathesis, platelet dysfunction, thrombocytopenia with platelet count <100,000/microliter, or documented coagulopathy
20. Significant alcohol consumption, defined as more than 2 drink units per day (equivalent to 20 g) in women and 3 drink units per day (equivalent to 30 g) in men, or inability to reliably quantify alcohol intake
21. Active substance abuse, based on Investigator judgment, including inhaled or injected drugs, within 1 year prior to the initial screening
22. Significant weight loss within the last 6 months (e.g., >10% total body weight loss)
23. Hepatic decompensation defined as the presence of any of the following:

    1. Serum albumin less than 3.5 g/dL
    2. International normalized ratio (INR) greater than 1.4 (unless due to therapeutic anticoagulants)
    3. Total bilirubin greater than 2 mg/dL with the exception of Gilbert syndrome
    4. History of esophageal varices, ascites, or hepatic encephalopathy
24. ALT or AST greater than 200 U/L
25. Diagnosis of liver cirrhosis
26. Chronic liver or biliary disease of the following etiology:

    1. History or diagnosis of Hepatitis B
    2. History or diagnosis of Hepatitis C
    3. History or diagnosis of current active autoimmune hepatitis
    4. History or diagnosis of primary biliary cholangitis (PBC)
    5. History or diagnosis of primary sclerosing cholangitis
    6. History or diagnosis of Wilson's disease
    7. History or diagnosis of alpha-1-antitrypsin deficiency
    8. History or diagnosis of hemochromatosis
    9. History or evidence of drug-induced liver disease, as defined on the basis of typical exposure and history
    10. Known bile duct obstruction
    11. Suspected or proven liver cancer
27. History of acute or chronic pancreatitis
28. Subjects unable to undergo CT for any reason
29. Currently enrolled in any other investigational trial
30. History of an acute neurologic event including epilepsy, seizures, stroke, and transient ischemic attack.
31. Iliac/femoral artery stenosis precluding insertion of the catheter
32. Human immunodeficiency virus (HIV)
33. Subjects with a history of adverse reaction to heparin or heparin induced thrombocytopenia (HIT)
34. Subjects with conditions that can affect RBC turnover, those who have received a blood transfusion in the past 90 days, or expect to have an elective procedure during the course of the study that may require blood transfusion
35. Not a candidate for surgery or general anesthesia
36. Unwilling to comply with study requirements, including medication run-in, SMBG, patient diary and follow-up visits
37. Subjects with implantable pacemakers, implantable cardiac defibrillators or implantable neurostimulators

    Anatomic Exclusions from CT Angiogram
38. Replaced or accessory LHA or RHA determined on CT angiogram.
39. Vessel tortuosity or variant vascular anatomy that could preclude the access or maneuvering of the device from the femoral artery to the target location
40. Evidence of CHA and/or portal vein intraluminal thrombus
41. CHA vessel diameter <4.0mm or >7.0mm
42. CHA diameter stenosis >30%
43. CHA vessel length <20mm

Ages: 22 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2020-07-28 (Actual); Primary Completion 2022-03-02 (Actual); Study Completion 2022-12-19 (Actual)

PRIMARY OUTCOMES:
Rate of Serious Adverse Device Effects | Index Procedure through 90 days
  The incidence rate of serious adverse device effects (SADEs) from time of Index Procedure through 90 days.

SECONDARY OUTCOMES:
Change in glycemic control: HbA1c | 30, 90, 180 and 365 days
  Change from baseline in glycemic control as indicated by HbA1c blood test
Change in glycemic control - FPG | 30, 90, 180 and 365 days
  Change from baseline in glycemic control as indicated by fasting plasma glucose blood test
Change in glycemic control - Insulin | 30, 90, 180 and 365 days
  Change from baseline in glycemic control as indicated by insulin blood test during Mixed Meal Tolerance Test
Change in glycemic control - C-peptide | 30, 90, 180 and 365 days
  Change from baseline in glycemic control as indicated by c-peptide blood test during Mixed Meal Tolerance Test
Change in office blood pressure | 30, 90, 180 and 365 days
  Change from baseline in office blood pressure: systolic and diastolic
Change in liver steatosis | 90 and 365 days
  Change from baseline in liver steatosis from baseline as measured using MRI-PDFF
Adverse Event rate 365 days | Consent through 365 days
  Adverse Event rate: Summary of all reported adverse events during the study

CONTACTS AND LOCATIONS:
Locations (8):
- United States (8):
  - Cardiology, P.C., Birmingham, Alabama
  - Stanford University Medical Center, Stanford, California
  - AdventHealth Translational Research Institute, Orlando, Florida
  - Prairie Education & Research Cooperative (PERC), Springfield, Illinois
  - Metropolitan Cardiology Consultants, Coon Rapids, Minnesota
  - South Oklahoma Heart Research, LLC, Oklahoma City, Oklahoma
  - UPMC Pinnacle, Harrisburg, Pennsylvania
  - Soltero Cardiovascular Research Center, Dallas, Texas

IPD SHARING:
Plan to Share IPD: No